CLINICAL TRIAL: NCT04699201
Title: Prevenció De L'Hèrnia Incisional Per Tròcar
Brief Title: Trocar Site Incisional Hernia Prevention
Acronym: PHIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Joan XXIII de Tarragona. (Other)
Collaborators: Institut de Diagnostic per la Imatge (Other); Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, Joan Ferreres i Serafini, MD, 3rd year resident, General Surgery, Hospital Universitari Joan XXIII de Tarragona.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 156/2020
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Incisional Hernia
Keywords: Incisional Hernia, Umbilical Trocar, Preventive mesh
MeSH Terms: conditions — Incisional Hernia | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: Bicentric Randomized Controlled Trial. 2 allocation groups, parallel. Single blind. Enrollment: consecutive cases Time Perspective: Prospective
Who Masked: Participant
Masking Description: The participant will not know if the umbilical incision has been close by standard technique or with the preventive mesh.
  Also the radiologists performing the ultrasounds after 12 months will not have the information of Prosthesis/Control patient allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prosthesis (Experimental): Firstly, a laparoscopic cholecystectomy is performed. After suturing the aponeurosis with a J needle and 0 Polydioxanone, a lightweight, large-pore mesh made of PVDF monofilament (polyvinylidene fluoride - DynaMesh-CICAT, FEC Textiltechnik, Germany) will be placed onlay, overlapping 2cm in all directions from the edge of the aponeurosis incision at the umbilical trocar site. The mesh will be fixed to the aponeurosis with cyanoacrylate glue (Glubran®, GEM, Viareggio, Italy).
  Interventions: Procedure: Hincisional hernia prevention by onlay prosthesis trocar closure; Procedure: laparoscopic cholecystectomy; Diagnostic Test: Abdominal ultrasound
- Control (Active Comparator): Firstly, a laparoscopic cholecystectomy is performed. Closure of the aponeurosis will be performed by standard procedure: under direct vision, suturing the aponeurosis with a J needle and 0 Polydioxanone, with a stitch interval of ≤ 5mm.
  Interventions: Procedure: laparoscopic cholecystectomy; Diagnostic Test: Abdominal ultrasound

INTERVENTIONS:
Procedure: Hincisional hernia prevention by onlay prosthesis trocar closure — Hincisional hernia prevention by onlay prosthesis trocar closure
  Arms: Prosthesis
Procedure: laparoscopic cholecystectomy — Laparoscopic cholecystectomy with or without common bile duct exploration
Diagnostic Test: Abdominal ultrasound — Ultrasound focused in abdominal wall defects on the trocar incisions, 12 months after the surgery

SUMMARY:
Objective: To test the preventive effect of the placement of an onlay mesh versus the use of a fascial closure device at the umbilical trocar site closure in order to prevent incisional hernia after laparoscopic surgery.

Methods: We designed a Two Center Randomized Controlled Trial were adult participants presenting for elective laparoscopic cholecystectomy, with or without an exploration of the common bile duct will be recruited, with allocation of each of them in 2 groups (prosthesis and control). Abdominal ultrasound scan focused on aponeurosis defects at the trocar sites will be performed at 12 postoperative months.

An ultrasound scan will be performed to avoid underdiagnosis bias since incisional hernia is frequently under detected by clinical examination.

Relevance: The prevalence of incisional hernia after laparoscopy might be as high as 30%, due to this reason is paramount to find a better closure technique.

There are few studies about incisional hernia including radiological exams in order to provide the exact prevalence of this pathology, even fewer literature exists about incisional hernia after laparoscopic procedures.

DETAILED DESCRIPTION:
OBJECTIVE To test the preventive effect of the placement of an onlay mesh at the time of umbilical trocar site closure in order to prevent incisional hernia after laparoscopic surgery.

The estimated prevalence of incisional hernia after laparoscopy is 15- 25%, being even higher among patients with risk factors. Many different closure techniques exist, however few of them have been tested in Randomised Control Trials. Most of them lack an image technique to provide more accurate results.

METHODOLOGY

We designed a Two Center, Randomized Controlled Trial that will enroll patients undergoing laparoscopic cholecystectomy, with or without an exploration of the common bile duct. Participants will be randomized to 2 groups. The pneumoperitoneum technique will be achieved by Hasson technique. The closure procedure will take place at the end of the surgery, after the cholecystectomy is performed:

* Prosthesis: after suturing the aponeurosis with a J needle and 0 Polydioxanone, a lightweight, large-pore mesh made of PVDF monofilament (polyvinylidene fluoride - DynaMesh-CICAT, FEC Textiltechnik, Germany) will be placed onlay, overlapping 2cm in all directions from the edge of the aponeurosis incision at the umbilical trocar site. The mesh will be fixed to the aponeurosis with cyanoacrylate glue (Glubran®, GEM, Viareggio, Italy).
* Control: Closure of the aponeurosis will be performed by standard procedure: under direct vision, suturing the aponeurosis with a J needle and 0 Polydioxanone, with a stitch interval of ≤ 5mm.

An abdominal ultrasound scan focused on aponeurosis defects at the trocar sites will be performed at 12 postoperative months. Minimum follow-up will be 12 months.

All the adverse events will be registered and classified according to the Clavien Dindo classification.

An ultrasound scan will be performed to avoid underdiagnosis bias since incisional hernia is frequently under detected by clinical examination.

Relevance: The prevalence of incisional hernia after laparoscopy might be as high as 30%, due to this reason is paramount to find a better closure technique.

There are few studies about incisional hernia including radiological exams in order to provide the exact prevalence of this pathology, even fewer literature exists about incisional hernia after laparoscopic procedures.

Univariate descriptive analysis will present the results as means (with standard deviation and range) for the continuous variables and as numbers and percentages for the categorical variables. Bivariate analysis will be carried out among the variables of interest to describe their level of correlation and evaluate the possible differences between them. To evaluate the differences between the continuous variables we will use the comparison of means based on the T-Student and for the comparison of categorical variables the Chi-square test. Finally, linear regression models and generalized linear models (as appropriate depending on the response variable) will be used to study the dependence of the variables of interest, with other factors of study. Statistical analysis will be carried out using the SPSS (Statistical Package for the Social Sciences) Software (IBM SPSS Statistics 23). All tests will be bilateral with a level of significance of 5%. 100% of the data recorded will be analyzed, and the proportion of values lost in the variables of interest will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic cholecystectomy, with or without an exploration of the common bile duct, undergoing surgery in our hospital
* ASA (American Society of Anesthesiologists) <IV

Exclusion Criteria:

* Allergy or intolerance to any of the mesh components
* Patients presenting already primary or incisional hernia of the abdominal wall
* ASA ≥IV
* Intraoperative conversion to laparotomy
* Emergency surgery
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of incisional hernia | 12 months
  The primary endpoint is the incidence of incisional hernia in the 2 groups. Because incisional hernia may occur within the first months after surgery, assessment will be carried out during scheduled clinical visits over 12 months. The presence of incisional hernia will be evaluated by physical examination and radiologically by an abdominal US scan performed at the end of follow-up (12 months after operation).

SECONDARY OUTCOMES:
Perioperative complications | 30 days
  Secondary endpoints will be perioperative complications, including wound infection, haematoma, pain and reoperation.
Economical impact | 12 months
  We will compare on one side the cost of the mesh and the glue and on the other side the costs of reoperation and hospital stay in case of appearance of incisional hernias.

CONTACTS AND LOCATIONS:
Overall Officials: Carles Olona Casas, MD, Study Director — Hospital Universitari de Tarragona
Locations (2):
- Spain (2):
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona, Tarragona
  - Pius, Hospital de Valls, Valls, Tarragona

IPD SHARING:
Plan to Share IPD: No